CLINICAL TRIAL: NCT06830863
Title: A Phase 1/2, Multicenter, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety, Bioavailability, and Effect of Topically Administered ATR04-484 for Moderate to Severe EGFRi-Associated Dermal Toxicity
Brief Title: A Study to Evaluate Topical ATR04-484 for EGFRi-Associated Dermal Toxicity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azitra Inc. (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATR04-EGFR-101
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: EGFR Inhibitor-associated Rash
Keywords: EGFR; acneiform; EGFR inhibitor-associated rash; EGFRi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATR04-484 (Experimental): Topically applied ATR04-484
  Interventions: Drug: ATR04-484
- Vehicle (Placebo Comparator): Topically applied vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ATR04-484 — ATR04-484 is a recombinant live biotherapeutic product (rLBP) containing the engineered S. epidermidis strain SE484 in an ointment formulation for topical use
  Other Names: ATR-04
  Arms: ATR04-484
Drug: Vehicle — Topically applied vehicle.
  Arms: Vehicle

SUMMARY:
The goal of this randomized clinical trial is to learn if topical treatment with ATR04-484 can treat skin rash in patients undergoing EGFR inhibitor (EGFRi) therapy. The primary goal of the study is to determine safety and tolerability of ATR04-484, and the secondary goal of the study is to assess efficacy signals of ATR04-484. Researchers will compare treatment of ATR04-484 to its vehicle. Participants will:

* Apply ATR04-484 or vehicle daily for 28 days
* Visit the clinic periodically for evaluation and sample collection

DETAILED DESCRIPTION:
This is a multicenter, randomized, blinded, vehicle-controlled Phase 1/2 trial of topically applied ATR04-484 in adult patients with moderate to severe EGFRi-related non-infected dermal toxicity affecting the face. The neck, chest, back, and other areas may also be affected.

The safety, bioavailability, pharmacodynamics (PD), and preliminary effect of ATR04-484 (at a single concentration) will be compared to that of its vehicle, in 2 patient cohorts. In each cohort, eligible patients will be randomized (3:1 ratio) to ATR04-484 or its vehicle. The initial cohort (n = 8) will receive a single 4 g application of the study drug to the face, chest, and back, followed by a 7-day observation period. Upon completion of this observation period, the patients in this cohort may continue in the study with daily applications of study drug for an additional 28 days. Following a safety observation period, a subsequent cohort (n = 24) may be enrolled and will receive a 4 g application of the study drug once daily for 28 days. Each cohort will be followed for 28 days after the last application of study drug.

Clinical assessments of treatment effect will be evaluated at each area that has received a full application of study drug (coverage of all lesional surfaces). The primary endpoint is safety and tolerability. Secondary endpoints including clinical efficacy, including: (1) the severity of the dermal toxicity using a 5-point regional assessment scale, based on modified CTCAE descriptors for skin toxicity (including a score of 0 for clear or unaffected skin through 4 for severely affected skin); (2) numeric rating scales for pruritus and pain; and (3) a quality-of-life assessment (Functional Assessment of Cancer Therapy-EGFRI 18 [FACT-EGFRI 18]). Bioavailability of ATR04-484 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Has Grade 2 or 3 non-infected moderate to severe EGFRi-related dermal toxicity affecting the face (the neck, chest, back and other areas may also be affected)

Exclusion Criteria:

* Significant skin disease other than EGFRi-related dermal toxicity
* Treatment with topical mid- to high-potency topical corticosteroids, or topical antibiotics or antibacterial washes on the face, neck, chest, or back within 14 days prior to baseline; treatment with systemic antibiotics or systemic corticosteroids within 14 days prior to baseline
* Residing with an immunocompromised person residing with them in the same dwelling from the baseline visit through 2 weeks after the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 57 days
  Treatment-emergent adverse events

SECONDARY OUTCOMES:
Severity of dermal toxicity | 57 days
  Investigator assessment of dermal toxicity using a 5-point regional assessment scale, based on modified CTCAE descriptors for skin toxicity (including a score of 0 for clear or unaffected skin through 4 for severely affected skin).
Pruritus | 57 days
  Patient reported via numeric rating scale for reflective (24 hour) pruritus
Quality-of-life assessment | 57 days
  Patient reported using Functional Assessment of Cancer Therapy-EGFRI 18 [FACT-EGFRI 18]

OTHER OUTCOMES:
Bioavailability of ATR04-484 | 57 days
  The bioavailability of SE484 will be assessed by qPCR

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - Yale University School of Medicine, New Haven, Connecticut
  - NYU Langone, New York, New York
  - The Ohio State University, Gahanna, Ohio
  - MD Anderson, Houston, Texas
  - Inova Schar Cancer, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No